CLINICAL TRIAL: NCT05235555
Title: Safety and Effectiveness of Transcatheter Aortic Valve Implantation - EffecTAVI Registry
Brief Title: EffecTAVI Registry
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Professor, Federico II University
Other Study IDs: 231/18
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Aortic Stenosis; Transcatheter Aortic Valve Replacement; TAVI
Keywords: Aortic Stenosis; Transcatheter Aortic Valve Replacement; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with symptomatic severe AS undergoing TAVI.
  Interventions: Device: Transcatheter heart valve (THV) with CE approval

INTERVENTIONS:
Device: Transcatheter heart valve (THV) with CE approval — TAVI trough femoral access or alternative routes

SUMMARY:
Aortic stenosis (AS) is the most common valvular heart disease among elderly population, with a increasing prevalence due to population ageing. In developed countries, the prevalence of severe AS among ≥75 years is approximately 3.4%. The onset of symptoms is associated with a poor prognosis. Indeed, mortality increases once symptoms appears.

For several decades, surgical aortic valve replacement (SAVR) has been the standard of care for symptomatic AS. Transcatheter aortic valve implantation (TAVI) was introduced as alternative treatment in inoperable patients in 2002. In the last two decades TAVI has led to a paradigm shift in the treatment of severe AS, representing a less invasive alternative to surgery. TAVI has shown to be non-inferior or superior to SAVR in several large-scale randomized clinical trials (RCTs) across the full spectrum of surgical risks. The newly available evidence has led to an expansion of guideline recommendations for TAVI. Furthermore, newer generations of transcatheter heart valve (THV) design, better patient selection, and technical enhancements have driven improvement in safety and reduction of procedural complications over time.

This observational study aim to prospectively evaluate the safety and efficacy of the procedure and clinical outcomes in patients undergoing TAVI.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is the most common valvular heart disease among elderly population, with a increasing prevalence due to population ageing. In developed countries, the prevalence of severe AS among ≥75 years is approximately 3.4%. The onset of symptoms is associated with a poor prognosis. Indeed, mortality increases once symptoms appears.

For several decades, surgical aortic valve replacement (SAVR) has been the standard of care for symptomatic AS. Transcatheter aortic valve implantation (TAVI) was introduced as alternative treatment in inoperable patients in 2002. In the last two decades TAVI has led to a paradigm shift in the treatment of severe AS, representing a less invasive alternative to surgery. TAVI has shown to be non-inferior or superior to SAVR in several large-scale randomized clinical trials (RCTs) across the full spectrum of surgical risks. The newly available evidence has led to an expansion of guideline recommendations for TAVI.

This observational study aim to prospectively evaluate the safety and efficacy of the procedure and clinical outcomes in patients undergoing TAVI.

EffectTAVI is an observational, monocentric registry promoted by Department of Advanced Biomedical Sciences of University of Naples Federico II.

The aim is to collect clinical, procedural, echocardiographic data and to evaluate the clinical outcomes of TAVI procedure.

Study population: consecutive patients with symptomatic severe AS candidate to TAVI, established by the multi-disciplinary Heart Team according to current guidelines recommendations.

Severe AS will be defined according to the following echocardiographic criteria:

* Aortic valve area: < 1 cm2
* Indexed aortic valve area: < 0,6 cm2/m2
* Mean aortic valve gradient: ≥ 40 mmHg
* Peak aortic jet velocity: ≥ 4,0 m/sec

TAVI can be performed using several arterial access: transfemoral, transapical, trans-subclavian and trans-aortic.

Written informed consent will be obtained for all patients for participation in this registry.

After hospital discharge, clinical follow-up will be performed at 30-day, 6 months and 1-year after TAVI. All adverse events were systematically collected and classified according to the definitions of the Valve Academic Research Consortium (VARC)-3 criteria.

Clinical, procedural and follow-up data will be anonymously entered in a web-based database RedCap (https://www.redcap.unina.it/redcap/). Patients will be entered with a pseudonym generated by the data collection system.

The pseudonym does not allow the identification of the patient and, therefore, meets the European criteria for the acquisition of data online.

The access to the online database is allowed through the use of a personal password, provided to the Primary Investigator and to the Co-Investigators involved in the study.

Data analysis will be performed by the investigators of the Department of Advanced Biomedical Sciences.

The extensive case studies that investigators expect to collect will be useful to establish clinical, procedural and follow-up data in short, medium and long term of patients with severe aortic stenosis undergoing TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic severe AS or degenerated bioprosthetic aortic valve and suitable for TAVI according to Heart Team evaluation;
2. Ability to provide informed consent.

Exclusion Criteria:

1. Contraindications to TAVI: e.g. evidence of intracardiac mass, thrombus or vegetation, endocarditis;
2. Poor adherence to scheduled follow-up;
3. Unable to understand and follow study-related instructions.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic severe AS candidate to TAVI, established by the multi-disciplinary Heart Team according to the current guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 30 days
  All cause mortality
All cause mortality | 1 year
  All cause mortality

SECONDARY OUTCOMES:
Cardiovascular mortality | 30 days
  Cardiovascular mortality
Cardiovascular mortality | 1 year
  Cardiovascular mortality
Number of participants with neurological events | 30 days
  Neurological events
Number of participants with neurological events | 1 year
  Neurological events
Number of participants with bleeding events | 30 days
  Bleeding events
Number of participants with bleeding events | 1 year
  Bleeding events
Vascular and access-related complications | 30 days
  Vascular and access-related complications
Vascular and access-related complications | 1 year
  Vascular and access-related complications
Number of participants with new conduction disturbances and arrhythmias | 30 days
  New conduction disturbances and arrhythmias
Number of participants with new conduction disturbances and arrhythmias | 1 year
  New conduction disturbances and arrhythmias
Number of participants with acute kidney injury | 30 days
  Acute kidney injury
Number of participants with acute kidney injury | 1 year
  Acute kidney injury
Number of participants with myocardial infarction | 30 days
  Myocardial infarction
Number of participants with myocardial infarction | 1 year
  Myocardial infarction
Hospitalization or re-hospitalization | 30 days
  Any admission after the index hospitalization or study enrolment to an inpatient unit or hospital ward for ≥24 h, including an emergency department stay.
Hospitalization or re-hospitalization | 1 year
  Any admission after the index hospitalization or study enrolment to an inpatient unit or hospital ward for ≥24 h, including an emergency department stay.
Cardiac structural complications | 30 days
  Any cardiac structure occurring during the procedure involving the aortic annulus, left ventricle outflow tract, ventricular septum, left or right ventricle, left or right atrium, mitral valve apparatus, tricuspid valve apparatus, coronary sinus, and pericardial effusion.
Cardiac structural complications | 1 year
  Any cardiac structure occurring during the procedure involving the aortic annulus, left ventricle outflow tract, ventricular septum, left or right ventricle, left or right atrium, mitral valve apparatus, tricuspid valve apparatus, coronary sinus, and pericardial effusion.
Number of participants with bioprosthetic valve dysfunction | 30 days
  Bioprosthetic valve dysfunction
Number of participants with bioprosthetic valve dysfunction | 1 year
  Bioprosthetic valve dysfunction
Number of participants with leaflet thickening | 30 days
  Hypo-attenuated leaflet thickening (HALT)
Number of participants with leaflet thickening | 1 year
  Hypo-attenuated leaflet thickening (HALT)
Number of participants with leaflet reduced motion | 30 days
  Reduced leaflet motion (RLM)
Number of participants with leaflet reduced motion | 1 year
  Reduced leaflet motion (RLM)
Number of participants with clinically significant valve thrombosis | 30 days
  Clinically significant valve thrombosis
Number of participants with clinically significant valve thrombosis | 1 year
  Clinically significant valve thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Esposito, MD, PhD, Principal Investigator — Federico II University
Locations (1):
- Federico II University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e35-e71. doi: 10.1161/CIR.0000000000000932. Epub 2020 Dec 17. PMID 33332149
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Leon MB, Mack MJ, Hahn RT, Thourani VH, Makkar R, Kodali SK, Alu MC, Madhavan MV, Chau KH, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Blanke P, Leipsic JA, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Herrmann HC, Szeto WY, Genereux P, Pershad A, Lu M, Webb JG, Smith CR, Pibarot P; PARTNER 3 Investigators. Outcomes 2 Years After Transcatheter Aortic Valve Replacement in Patients at Low Surgical Risk. J Am Coll Cardiol. 2021 Mar 9;77(9):1149-1161. doi: 10.1016/j.jacc.2020.12.052. PMID 33663731
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579